CLINICAL TRIAL: NCT04237740
Title: Evaluation of the Efficacy and Safety of Relenvatinib in the Tatment of Recurrence of Hepatocellular Carcinoma After Liver Transplantation: a One-arm, Open-label Study
Brief Title: Relenvatinib in the Tatment of Recurrence of Hepatocellular Carcinoma After Liver Transplantation
Acronym: RRHCCLT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Renji8790
Record Dates: First submitted 2020-01-19; First posted 2020-01-23 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Hepatocellular Carcinoma; Liver Transplantation
Keywords: recurrent hepatocellular carcinoma; liver transplantation; relenvatinib
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: The cases are from patients with recurrent hepatocellular carcinoma who underwent liver transplantation in the liver surgery department of Shanghai Renji Hospital. The enrolled patients are treated with lenvatinib (dose: body weight < 60 kg: 8 mg/day, body weight ≥ 60 kg 12 mg/day).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- relenvatinib (Experimental): The enrolled patients are treated with lenvatinib (dose: body weight < 60 kg: 8 mg/day, body weight ≥ 60 kg 12 mg/day).
  Interventions: Drug: relenvatinib

INTERVENTIONS:
Drug: relenvatinib — The enrolled patients are treated with lenvatinib (dose: body weight < 60 kg: 8 mg/day, body weight ≥ 60 kg 12 mg/day).
  Other Names: relenvatinib treatment

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of lenvatinib in the treatment of recurrence of hepatocellular carcinoma after liver transplantation.

DETAILED DESCRIPTION:
The research is an open, one-arm, single-center study. 40 patients with recurrence of hepatocellular carcinoma after liver transplantation are included according to the criteria of admission. The enrolled patients are treated with lenvatinib (dose: body weight < 60 kg: 8 mg/day, body weight ≥ 60 kg 12 mg/day). The baseline data of patients are collected before allocation. Serum and imaging examination are checked regularly every month to monitor the recurrence of hepatocellular carcinoma and the side effects of lenvatinib. The efficacy and safety of lenvatinib in the treatment of recurrence of hepatocellular carcinoma are observed, and the clinicopathological factors affecting the efficacy of lenvatinib are analyzed. When side effects of lenvatinib occur, the dosage can be reduced according to the patients' condition until discontinuation. When tumor advances, a multidisciplinary team will draw up specific treatment plans according to the patients' condition.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are with recurrence of hepatocellular carcinoma after liver transplantation who are unfit for or reject the treatment of hepatectomy, retransplantation, local therapy (radiofrequency ablation, interventional therapy, radiotherapy) and chemotherapy.
2. aged 18 to 75.
3. ECOG physical condition was 0-2 points.
4. Child-Pugh A grade of liver function.
5. Targeted therapy is acceptable within 1-2 months after liver transplantation.
6. Immunosuppressive regimen consists of calcineurin inhibitor, mycophenolate mofetil and sirolimus.
7. No history of surgical resection of liver tumors and targeted drug therapy before liver transplantation.
8. Good liver, kidney and bone marrow function: or PT within 6 seconds over normal upper limit.
9. For fertile female patients, the serum/urine pregnancy test should be negative within 7 days before treatment.
10. All male and female participants must take reliable contraceptive measures during the trial and within four weeks after the end of the trial.

12.The participants have the capability of oral medication. 13.The participants must sign the consent form.

Exclusion Criteria:

1. Patients are with other malignant tumors simultaneously.
2. Patients are anaphylaxis to the inactive ingredients of lenvatinib or drugs.
3. Pregnant or lactating women (Female participants need pregnancy test within 7 days before treatment).
4. Preoperative history of severe cardiovascular disease: congestive heart failure > NYHA grade 2; active coronary heart disease (myocardial infarction occurred within 6 months before entry into the study); severe arrhythmia requiring antiarrhythmic treatment (allowable use of beta-blockers or digoxin); uncontrolled hypertension.
5. History of HIV infection.
6. Severe clinical active infections
7. Epilepsy patients requires medication (e.g. steroids or antiepileptic drugs).
8. Patients with kidney diseases requires renal dialysis.
9. Drug abuse, medical symptoms, mental illness or social status that may interfere with participants'participation in research or evaluation of research results.
10. Patients who could not swallow oral drugs, such as those with severe upper gastrointestinal obstruction and need gastric tube feeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
3 years recurrence-free survival rate | 3 years
  Tumor recurrence within 3 years

SECONDARY OUTCOMES:
1 year recurrence-free survival rate | 1 year
  Tumor recurrence within 1 year
5 years recurrence-free survival rate | 5 years
  Tumor recurrence within 5 years
1 year overall survival rate | 1 year
  overall survival with one year
3 years overall survival rate | 3 years
  overall survival with 35 years
5 years overall survival rate | 5 years
  overall survival with 5 years

CONTACTS AND LOCATIONS:
Overall Officials: qiang xia, doctor, Study Chair — RenJi Hospital

IPD SHARING:
Plan to Share IPD: No